CLINICAL TRIAL: NCT02570607
Title: Relevance of Preoperative BNP as a Biomarker of Postoperative Cardiovascular Complications in Major Non-cardiac Adult Surgery
Brief Title: Preoperative BNP as Biomarker of Postoperative Cardiovascular Complications
Acronym: BNP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 15-PP-10
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Postoperative Cardiovascular Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: BNP dosage

SUMMARY:
BNP is a hormone that predicts preoperatively the occurrence of postoperative cardiovascular complications. In practice, the problem is that the practitioner don't know the most opportune moment for the preoperative sample or what threshold used to classify our patient in patients at risk of cardiovascular complication or not at risk.

The purpose of this study is to determine the best time to dose the preoperative BNP with a specific threshold being associated with it allowing the practitioner to assess more accurately the post operative cardiovascular risk patients and possibly offer them strategies taking different load.

The BNP will be dosed during the anesthetic consultation and the day of surgery in immediate preoperative operating room. Post-operative cardiovascular complications will be collected during hospitalization of the patient and by telephone contact on the 28th day, 90th day and 6th postoperative months.

The investigator then establish the threshold BNP most informative for both sampling times and then compare them to determine the most discriminating dosage and thus the most appropriate time for the determination of BNP.

DETAILED DESCRIPTION:
The morbidity and mortality of non-cardiac major surgery is mainly due to cardiovascular complications. BNP is a hormone for predicting preoperatively the occurrence of these complications. Widely used in cardiac surgery, it is not routinely used in non-cardiac major surgery. His interest in this type of surgery has yet been proven by numerous studies.

In practice, the problem with this biomarker is the pratitioner do not know the most opportune moment for the preoperative dose or what threshold used to classify our patient patients at risk of cardiovascular complication or not at risk.

Indeed, recent literature reviews are used to highlight the fact that existing studies on the subject using each method or BNP assay devices and heterogeneous preoperative dosing of different times or even BNP not exactly specified. It thus appears as many different levels of BNP. Practitioners did not then know when dosing the BNP and what threshold is based.

The purpose of this study is to determine the best time to dose the preoperative BNP with a specific threshold being associated with it allowing the practitioner to assess more accurately the post operative cardiovascular risk patients and possibly offer them strategies taking different load.

The BNP will be dosed during the anesthetic consultation and the day of surgery in immediate preoperative operating room. Post-operative cardiovascular complications will be collected during hospitalization of the patient and by telephone contact on the 28th day, 90th day and 6th postoperative months.

The investigator then establish the threshold BNP most informative for both sampling times and then compare them to determine the most discriminating dosage and thus the most appropriate time for the determination of BNP.

There will be no immediate benefit to the patient but our study will help in the future, to adapt the management of perioperative patients depending on the value of pre immediate operative BNP to reduce postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Major patients who was not opposed to one additional sample

  * Who have to undergoing moderate or high cardiovascular risk non-ambulatory scheduled surgery with the exception of cardiac surgery
  * With predictable delay between the preoperative evaluation and the surgery > 15 days

Exclusion Criteria:

* Moderate cardiovascular risk surgeries (1-5%):
* Carotid Endarterectomy
* Surgery of the Head and Neck
* Thoracic surgery and intraperitoneal (thromboembolism)
* Orthopaedic surgery (thromboembolism)
* Prostate Surgery (thromboembolism)

High cardiovascular risk surgeries (> 5%):

* Aortic surgery with risk of sudden changes in blood pressure during clamping (acute pulmonary edema, ischemia)
* declamping (coronary perfusion)
* other major vascular surgery - peripheral vascular surgery - long surgery with significant blood loss or fluid and electrolyte

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient Who have to undergoing moderate or high cardiovascular risk non-ambulatory scheduled surgery with the exception of cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
occurrence of a complication or cardiovascular events | 2 years
  The endpoint is the occurrence of a complication or cardiovascular events (composite endpoint). A cardiovascular event is defined by the occurrence of syndromes such as IDM, acute cardiogenic lung edema, a rhythm disturbance (ACFA, flutter, TV, FV) or c